CLINICAL TRIAL: NCT02422368
Title: The Effect of a New Antioxidant Combination (ASTED) on Moderate to Severe Thyroid Eye Disease, a Double Blind Placebo Controlled Randomized Clinical Trial
Brief Title: The Effect of a New Antioxidant Combination (ASTED) on Moderate to Severe Thyroid Eye Disease
Status: Withdrawn | Phase: Phase 2 / Phase 3 | Type: Interventional
Why Stopped: Do not access to the drug
Sponsor: Iran University of Medical Sciences (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 93-02-124-24581
Record Dates: First submitted 2015-04-11; First posted 2015-04-21 (Estimated); Last update posted 2022-01-10 (Actual); Status verified 2021-01

CONDITIONS: Thyroid Eye Disease
Keywords: Graves' ophthalmopathy; Antioxidant; Activity; Severity
MeSH Terms: conditions — Graves Ophthalmopathy; Motor Activity | interventions — Methylprednisolone

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Methylprednisolone + ASTED (Experimental): ASTED (Antioxidant Supplements for Thyroid Eye Disease) includes : B-Carotene (6 mg)+ Vit.C (200 mg) + Vit.E (200 mg) + Nicotinamide(20mg) + Selenium(200mic.) + Zinc oxide (8 mg) + Copper gluconate or oxide (1mg) + Manganese chloride (1.8 mg), Twice a day for 6 months
  Methylprednisolone includes :
  Methylprednisolone tablet of 50 and 5 mg, company….) 1mg/kg for the first 2 weeks, 0.8mg/kg for 2 weeks, 0.7 mg/kg for 2 weeks, and then tapering off the methylprednisolone in 6 weeks (total duration of 12 weeks) by 8-10 mg per week. For example, a patient with 75 kg weight will receive 75 mg for 2 weeks, 60 mg for 2 weeks, 52.5 mg for 2 weeks, and then decreasing by 8-10 mg per week for 6 weeks. The dose regiment will be written and handed to the patient on the first visit and will be monitored during the follow up.
  Interventions: Drug: Methylprednisolone + ASTED
- Methylprednisolone + Placebo (Placebo Comparator): Placebo Twice a day for 6 months Methylprednisolone prescribes as the same as arm 1
  Interventions: Drug: Methylprednisolone +Placebo

INTERVENTIONS:
Drug: Methylprednisolone + ASTED — ASTED tablet: Twice daily for 6 months
  Methylprednisolone:
  Methylprednisolone tablet of 50 and 5 mg, company….) 1mg/kg for the first 2 weeks, 0.8mg/kg for 2 weeks, 0.7 mg/kg for 2 weeks, and then tapering off the methylprednisolone in 6 weeks (total duration of 12 weeks) by 8-10 mg per week. For example, a patient with 75 kg weight will receive 75 mg for 2 weeks, 60 mg for 2 weeks, 52.5 mg for 2 weeks, and then decreasing by 8-10 mg per week for 6 weeks. The dose regiment will be written and handed to the patient on the first visit and will be monitored during the follow ups.
  Arms: Methylprednisolone + ASTED
Drug: Methylprednisolone +Placebo — Placebo: twice daily
  Methylprednisolone:
  Methylprednisolone tablet of 50 and 5 mg, company….) 1mg/kg for the first 2 weeks, 0.8mg/kg for 2 weeks, 0.7 mg/kg for 2 weeks, and then tapering off the methylprednisolone in 6 weeks (total duration of 12 weeks) by 8-10 mg per week. For example, a patient with 75 kg weight will receive 75 mg for 2 weeks, 60 mg for 2 weeks, 52.5 mg for 2 weeks, and then decreasing by 8-10 mg per week for 6 weeks. The dose regiment will be written and handed to the patient on the first visit and will be monitored during the follow ups.
  Arms: Methylprednisolone + Placebo

SUMMARY:
ASTED (Antioxidant Supplements for TED) trial is an investigator-initiated, randomized, triple masked, clinical trial of a selected combination of vitamins and minerals versus placebo in patients with moderate to severe thyroid eye disease. The trial has a parallel-arm design.

DETAILED DESCRIPTION:
Primary aim: To investigate if ASTED or as compared with placebo could affect the course of TED either by enhancing improvement or preventing worsening in patients with Moderate to severe TED thyroid eye disease (TED) based on:

1. Total eye score (NOSPECS severity score) 1 Total eye score is used to assess the severity of TED, which was calculated by multiplying each class of the NOSPECS system1 (except class 0) to its grade of severity (0-3), yielding a maximum total score of 63 and a minimum total score of 0 (the higher the number the worse the severity) The overall ophthalmic outcome is a composite score based on multiple items (Soft tissue, retraction, proptosis, diplopia, and corneal involvement); the use of a composite score circumvents the problem arising from the presence of improvement in one item and simultaneous worsening in another item.

   The severity score in each of the classes 1, 2, 3, and 4 will also be separately compared to evaluate the effect of different treatments on each sign.
2. Score of thyroid eye disease Quality of life questionnaire (TED-QOL) 2.

Secondary outcomes measures:

To compare possible change in:

1. Clinical activity score (CAS Score) 3 (7 items are scored in the beginning and 10 items are scored at 3 and 6 months)
2. Serum thyroid auto-antibodies (Anti-thyroid peroxidase (TPO), Anti-thyroglobulin) at 0, 3 and 6 months. Thyroid function test (Free T4, T3, and TSH) will be measured in all 3 visits0
3. Side effects

ELIGIBILITY:
Inclusion Criteria:

* Moderate to severe TED of less than 18 months duration:
* Active state (Clinical activity score of 3 and more).
* No steroid and or any supplement treatment for the last 6 months.
* Euthyroidism
* Age 18-70 years.

Exclusion Criteria:

* Sight-threatening TED
* Pregnancy
* Drug and/or alcohol abuse
* Severe concomitant illness
* Inability to comply with the study protocol
* No informed consent
* Developing more severe TED (Sight threatening TED) in the course of the trial.
* Contraindications of steroid treatment.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2022-09-01 (Estimated); Primary Completion 2024-06 (Estimated); Study Completion 2024-11 (Estimated)

PRIMARY OUTCOMES:
Mean of total eye score changes (using NOSPECS severity score) | baseline, 1 month, 3 months, 6 months
  Total eye score change during study
Mean of "thyroid eye disease Quality of life" score changes (Using TED-QOL) | baseline, 1 month, 3 months, 6 months
  Changing quality of life during study period

SECONDARY OUTCOMES:
Mean of clinical activity score changes (CAS Score) | baseline, 1 month, 3 months, 6 months
  Change of clinical activity score during study period
Changes of serum thyroid auto-antibodies (Anti-thyroid peroxidase (TPO), Anti-thyroglobulin) | baseline, 1 month, 3 months, 6 months
  Change of serum thyroid auto-antibodies during study period
Changes of thyroid function test (Free T4, T3, and TSH) Levels | baseline, 1 month, 3 months, 6 months
  Change of thyroid function test during study period

CONTACTS AND LOCATIONS:
Overall Officials: Mohsen B Kashkouli, MD, Principal Investigator — IUMS
Locations (2):
- Iran (2):
  - Private Thyroid eye disease clinic, Tehran
  - Rassoul Akram Hospital, Tehran